CLINICAL TRIAL: NCT05726526
Title: A Pragmatic Randomized Controlled Trial of a CKD Specific Telemonitoring Platform to Minimize Adverse Outcomes in High Risk CKD Patients
Brief Title: CKD Specific Telemonitoring Platform to Minimize Adverse Outcomes in High Risk CKD Patients
Acronym: VIEWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Claudio Rigatto, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HS25046 (B2021:066)
Record Dates: First submitted 2021-08-16; First posted 2023-02-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease Stage 5; End Stage Renal Disease
Keywords: telemonitoring; chronic kidney disease; suboptimal dialysis initiation; digital health
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly allocated to the intervention group (usual care + the VIEWER virtual care platform) or the control group (usual care).
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention, patients and care providers will not be blinded; outcome assessment and statistical analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will be provided with a wireless BP cuff, weight scale, transcutaneous O2 sat monitor, wearable motion tracker and mobile tablet with the VIEWER application. Patients will be trained to use the VIEWER platform either virtually or in person. Patients will be guided through a daily self-assessment routine via the app (BP, weight, O2 saturation, step count upload) and weekly ESAS-r survey. Participants will use the VIEWER platform for 12 months ( or until dialysis initiation) in addition to receiving usual care. Additionally, participants will complete the UK Kidney PREM score (adapted to CKD) and the Health related QOL using KDQOL-SF via REDCap or paper form at baseline, 3, 6, 9 and 12 months (or every 3 months until dialysis initiation), and the System Usability Scale (SUS) at 12 months.
  Interventions: Device: VIEWER virtual care platform
- Control Group (No Intervention): Participants randomized to the control group will continue to receive usual care either virtually via telephone or video call or in person depending on COVID-19 restrictions in place. Participants will complete the UK Kidney PREM score (adapted to CKD) and the Health related QOL using KDQOL-SF via REDCap or paper form at baseline, 3, 6, 9 and 12 months (or every 3 months until dialysis initiation).

INTERVENTIONS:
Device: VIEWER virtual care platform — VIEWER is a tablet based, CKD specific home telemonitoring platform developed by our team of patients and researchers that integrates data from a wireless blood pressure cuff, weigh scale, transcutaneous O2 sat monitor and wearable motion tracker via a tablet and custom app.
  Arms: Intervention Group

SUMMARY:
The main purpose of this trial is to determine whether the addition of the VIEWER virtual care platform to usual care will lead to a reduction in composite emergency department (ED) visits and/or hospitalizations/or increase the perceived safety of virtual care among patients and providers.

DETAILED DESCRIPTION:
Background: Chronic Kidney Disease (CKD) is an increasingly prevalent condition that represents a major national public health burden. The health transition from advanced CKD to the start of dialysis is a period of heightened vulnerability for many patients. Our data has demonstrated that during the 30-day period before the start of dialysis, there is a 10-fold increase in Emergency Department (ED) visits and hospitalizations related to kidney failure and its complications. Importantly, this spike occurs despite patients having frequent contact with their nephrology healthcare teams. For stable CKD patients, virtual monitoring could facilitate the communication of accurate and reliable data between patients and providers helping to avoid unnecessary ED visits and facilitate more optimal dialysis starts.

Design& Method: The VIEWER study is a national, pragmatic, multicenter randomized controlled trial across 5 Canadian sites from two provinces including:

1. Seven Oaks General Hospital (SOGH), Winnipeg, Manitoba.
2. St. Boniface hospital (SBH), Winnipeg, Manitoba.
3. Health Sciences center (HSC), Winnipeg, Manitoba.
4. Health Sciences Center, London, Ontario.
5. Scarborough Health Network (SHN), Scarborough, Ontario.

VIEWER is a CKD-specific virtual care platform that integrates data from a wireless Blood Pressure (BP) cuff, weight scale, transcutaneous O2 sat monitor, and wearable motion tracker. The patient-facing component of VIEWER (patient portal), is a custom application based on a mobile tablet that guides patients through a daily self-assessment routine using the connected devices. BP measurements, weight and oxygenation (as surrogates of volume status), and step counts (as a surrogate of functional status), provide semi-continuous longitudinal data on patient physical status. Additionally, patients are prompted to fill out a weekly symptom survey (Edmonton Symptom Assessment Score- revised; ESAS-r), a validated instrument of kidney failure symptoms. Patient data and ESAS scores are automatically uploaded to fully PHIA/HIPPA compliant servers where they are made available to the patients' care team through a secure, web-based provider portal. Provider notifications (flags) are generated for out-of-range values (i.e. BP, weights for volume management) and a secure messaging component allows for direct patient-provider communication. Participants will be trained to use the VIEWER platform by a member of the research team. On the provider side, two members of the care team at each site will be trained as "superusers" of the provider portal. These users will check and respond as needed daily (Monday to Friday) for flags and patient messages, and will respond or communicate as needed to the health care team as per local clinic standard operating procedures. Trends in measurements will be reviewed at multidisciplinary team rounds, which typically occur weekly. During routine clinic visits, trends in all objective and subjective measures will be available to review to inform clinical decision making. Consistent with our pragmatic design, we will not be proscriptive in how monitoring data are interpreted; rather, we ask that care teams consider this enriched data stream and incorporate that information according to their own protocols and clinical judgement.

Patients randomized to the control group will see their multidisciplinary CKD care teams as per usual care.

Follow-up visits and Focus Groups (or individual interview): Patient Reported Experience Measures (PREM) and Kidney Disease Quality of Life-Short Form (KDQOL-SF) will be measured at baseline, 3, 6, 9 and 12 months in all paticipanats. Usability, acceptability, and patient and provider perspective on the intervention will be assessed at the end of the trial using the System Usability Scale (SUS). In addition, two virtual focus groups will be conducted at the end of the study with a subset of participants and healthcare providers who used the VIEWER platform.

Statistical Methods:The primary outcome (time to first hospitalization or ED visit, censoring at dialysis or death) will be assessed using univariate Cox proportional hazards models and a Kaplan-Meier analysis with a log-rank test, as will the secondary outcomes of all-cause mortality, ED visits, hospitalization, and acute inpatient dialysis initiation. Change in overall PREM, KDQOL-SF and SUS scores will be assessed with two-sided t-test or Wilcoxon Rank Sum test as distributionally appropriate, and interpreted relative to their minimal important differences. All outcomes will be assessed at a two-sided alpha= 0.05. Subgroup analyses will be prespecified and limited to 1) eGFR greater or less than 10ml/min, 2) sex and gender (described below) 3) diabetes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Patient or primary caregiver can read and speak English
* Patient or patients substitute decision maker is able to provide informed consent
* Patient or primary care giver cognitively and physically capable and willing to use the VIEWER mobile application and perform self-measurements (i.e. weight, BP, etc.)
* Have stage 5 CKD (2 measurements of eGFR <15ml/min/1.73m2); eGFR will be calculated with the CKD-EPI equation, or have >40% chance of beginning dialysis in the next 2 years based on the Kidney Failure Risk Equation
* Followed in a multidisciplinary CKD clinic

Exclusion Criteria:

* Inability of self or caregiver assisted self-monitoring using VIEWER

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Composite of first hospitalization or emergency department (ED) visit | 12 months or until dialysis initiation
  It's defined as an inpatient admission to hospital or a visit to the emergency department, whatever is first". So, we will compare the time of the first hospital admission /and or ED visit between two groups.

SECONDARY OUTCOMES:
All-cause mortality | 12 months or until dialysis initiation
  The mortality rate will be compared between the intervention and control group.
Proportion of patients who have an acute inpatient initiation of dialysis. | 12 months or until dialysis initiation
  the rate of patients who started dialysis in the intervention and control groups during 1 year of follow-up.
Frequency of Emergency Department Visit | 12 months or until dialysis initiation
  The average frequency of ED visit will be compared in two study groups.
Frequency of formal clinic visits | 12 months or until dialysis initiation
  The average frequency of formal clinic visits will be compared between two study groups
UK Kidney PREM score (adapted to CKD) | baseline, 3, 6, 9 and 12 months (or every 3 months until dialysis initiation)
  The UK Kidney Patient Reported Experience Measure is a validated, self-reported scale that focuses on how kidney patients experience care. The UK Kidney PREM used for this trial consists of questions abstracted from the 2019 Kidney PREM. Possible scores range from 1 (strongly disagree) to 10 (strongly agree). The average total scores will be compared between intervention and control group.
Health related QOL using KQOL-SF | baseline, 3,6,9 and 12 months (or every 3 months until dialysis initiation)
  Kidney Disease Quality of Life- Short Form is a self-reported measure developed for individuals with kidney disease and those on dialysis. It includes 43 kidney disease targeted items, and 36 items that provide a measure of physical and mental health and 1 overall health rating item ranging from 0 (worst possible health) to 10 (best possible health).The average total scores will be compared between intervention and control groups.
System Usability Scale (SUS) | 12 months ( or at the time of dialysis initiation)
  The System Usability Scale measures the usability of a wide range of products and services including hardware and software. It consists of a 10 item questionnaire with 5 response options ranging from 1 (strongly disagree) to 5 (strongly agree). This will be assessed via focus groups held with a subset of patients.
Provider Perspectives towards intervention (qualitative) focus groups | 12 months (or end of study)
  Assessed via focus groups held with a subset of providers
Patient Perspectives towards intervention (qualitative) focus groups (or individual interview) | 12 months (or end of study)
  Assessed via focus groups held with a subset of patients
Proportion of patients greater than 80% adherence | 12 months (or end of study)
  tracked via VIEWER app

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Rigatto, MD, Principal Investigator — University of Manitoba
Locations (5):
- Canada (5):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Chronic Disease Innovation Centre, Seven Oaks Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Scarborough Health Network - General Hospital, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solati Z, Komenda P, Tangri N, Saul S, Bohm C, Ferguson T, Hager D, Barr B, Mysore P, Hougen I, Meraz-Munoz A, Jain AK, Tam P, Rigatto C. A Pragmatic Randomized Controlled Trial of a CKD-Specific Virtual Monitoring Platform to Minimize Adverse Outcomes in High-Risk CKD Patients: A Clinical Research Protocol. Can J Kidney Health Dis. 2025 Oct 5;12:20543581251359736. doi: 10.1177/20543581251359736. eCollection 2025. PMID 41058978